CLINICAL TRIAL: NCT01626040
Title: Evaluation of One-day Polyethylene Glycol Powder Solution for Colonoscopy in Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Petar Mamula, Medical Doctor, Children's Hospital of Philadelphia
Other Study IDs: 12-008643
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Water-Electrolyte Imbalance
MeSH Terms: conditions — Water-Electrolyte Imbalance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: No biospecimens are to be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEG-P prep: Children taking the one day polyethylene glycol powder preparation for outpatient colonoscopy
  Interventions: Drug: polyethylene glycol powder

INTERVENTIONS:
Drug: polyethylene glycol powder — A single group of children taking a polyethylene glycol powder preparation, dosage determined by patient weight, taken in one dose the day before colonoscopy

SUMMARY:
The purpose of this study is to examine the effects of current standard of care Polyethylene Gylcol powder (PEG-P)colonoscopy preparation on a patient's serum electrolytes, tolerance of the prep, and how well the bowel is cleansed. The primary aim is to determine the proportion of patients with clinically significant serum electrolyte abnormalities at the time of colonoscopy and how well the prep is tolerated. Secondary objectives include: 1) how well the bowel is cleansed with this preparation, and 2) to determine the most effective way to communicate instructions about the bowel preparation with the child and family.

DETAILED DESCRIPTION:
Design is prospective, descriptive observational study involving a single clinical encounter in the Endoscopy suite at CHOP Main at the time of colonoscopy. Patients prescribed the standard of care dosage for PEG-P by their primary gastroenterologist are considered for this study. Study procedures include collection of data from patients that are prescribed the PEG-P dose. In order to evaluate the safety, tolerability, and adherence to PEG-P bowel preparation, data collections include the following: review of medical records, tracking of communication from subjects/parents, blood draw, questionnaire and quality of prep will be assessed. Questionnaire results will be obtained at the initial and only visit. Patients will be given a questionnaire prior to colonoscopy to rate symptoms, ease of preparation and to rate the effectiveness of communication about the preparation. On the day of colonoscopy, prior to the procedure, patients will have an IV placed per standard procedure. At the time of IV placement, a basic metabolic panel and serum magnesium and phosphorus levels will be drawn through the IV for assessment of electrolyte abnormalities. Serum glucose will be captured from medical records as this is collected with standard of care. Patient/parents will grade the preparation tolerance filling out a questionnaire prior to colonoscopy. During colonoscopy, the endoscopist will grade the quality of preparation on a validated residual stool survey (Aronchick scale).

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 1 - 18 years
* patients receiving standard of care dosing for polyethylene glycol powder
* patients who had electrolyte results within the last 60 days of enrollment
* parental / guardian permission (informed consent)

Exclusion Criteria:

* Patients on the GI inpatient or consult service
* Weight less than 10 kg
* Pregnant or lactating females
* Non-English speaking patient or parent
* 5) Parents/guardians or subjects who, in the opinion of the Investigator/Study team, may be non-compliant with study schedules or procedures

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children undergoing outpatient colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2012-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
electrolyte disturbances | at the time of colonoscopy
  the proportion of patients with clinically significant serum electrolyte abnormalities at the time of colonoscopy
PEG-P preparation tolerance | at the time of colonoscopy
  Responses to a questionnaire regarding the tolerance of the PEG-P prep will be recorded

SECONDARY OUTCOMES:
Colonoscopy preparation efficacy | at the time of colonoscopy
  To assess the proportion of patients that have excellent or good quality preparation as scored by a validated residual stool survey called the Aronchick scale
Effective communication | at the time of colonoscopy
  Effectiveness of communication strategy about the prep and availability of staff to address questions reported by parents will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Petar Mamula, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States